CLINICAL TRIAL: NCT01932645
Title: Modern Genetic Methods to Test EPS Samples in Prostatitis Patients
Brief Title: Etiology Study of Prostatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Other Study IDs: H13-01947
Record Dates: First submitted 2013-08-08; First posted 2013-08-30 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Prostatitis
Keywords: prostatitis; pelvic pain; urinary symptoms; sexual dysfunction
MeSH Terms: conditions — Prostatitis; Pelvic Pain; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will have a digital rectal exam (DRE) performed and have their Expressed Prostatic Secretions (EPS) sampled as well as the first void after the DRE (other wise called the VB3 sample). Patients will also have their maximum urinary flow rate tested by voiding into a special machine. This will be done at the urology clinic, 6th floor Diamond Building.
  These biological samples will be tested for bacterial DNA rather than the traditional microbiological culturing techniques. Identification of these bacterial DNA will then be assessed between the groups to determine if prostatitis patients, in fact, do have more bacteria than normal controls.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prostatitis patients: We will enroll patients from the outpatient clinic who are suffering from pelvic pain (perineal, suprapubic, testicular, penile etc), have urinary symptoms and sexual dysfunction (primarily pain associated with ejaculation). Patients with these symptoms and identified as having prostatitis will be approached to enroll.
- Controls: Male patients seen in the outpatient clinic who do not have prostatitis (not suffering from pelvic pain (perineal, suprapubic, testicular, penile etc), and do not have urinary symptoms and sexual dysfunction (primarily pain associated with ejaculation)) will be approached to enrol as controls.

SUMMARY:
Prostatitis is so widespread a disease that affects people from youths to seniors, with approximately a third experiencing a remission of symptoms over a year follow-up. Although the etiology of prostatitis is still not clear, it is mainly thought to be due to infection of bacteria or other microorganisms. Up to now, there is still no research being done on the microbiome (bacterial species) of the prostate. The objective of this study is to look at the etiology of chronic prostatitis(bacteria or non-bacteria prostatitis), mainly focusing on the effect of bacteria in the prostate.

DETAILED DESCRIPTION:
Prostatitis is so widespread a disease that affects people from youths to seniors, with approximately a third experiencing a remission of symptoms over a year follow-up. Although the etiology of prostatitis is still not clear, it is mainly thought to be due to infection of bacteria or other microorganisms. Traditional techniques to identify bacteria (e.g. on agar petri plates) are limited in what they can identify. Although HMP (Human Microbiome Project) has turned many mysteries into common sense, little is done on the relationship of bacteria in the prostate for prostatitis. Up to now, there is still no research being done on the microbiome (bacterial species) of the prostate. The objective of this study is to look at the etiology of chronic prostatitis (bacteria or non-bacteria prostatitis), mainly focusing on the effect of bacteria in the prostate. Modern sequencing methods, such as 16s rRNA amplification, cloning and sequencing will be used to evaluate the role of bacteria in prostatitis. The basic idea is to survey the microbes present in expressed prostatic fluid using 16s sequencing to compare healthy men and prostatitis patients in a small cohort to see if there are correlations between microbes found and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* chronic prostatitis (bacteria or non-bacterial prostatitis) with pelvic pain and LUTS (low urinary tract symptom); diagnosed mainly by NIH-CPSI score. We use NIH-CPSI score 15 as a base line for identifying prostatitis patients:those scored more than 15 will be grouped as prostatitis patients.

Exclusion Criteria:

* Inadequate follow-up data
* Other types of prostatits patients
* Patients who in the opinion of the investigators would not be suitable for study
* UTI patients (within 6 months before enrolment)
* Antibiotics (within 6 months before enrolment)
* Urinary tract surgery (within 6 months before enrolment)

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with prostatitis (who are suffering from pelvic pain (perineal, suprapubic, testicular, penile etc), have urinary symptoms and sexual dysfunction (primarily pain associated with ejaculation)) vs controls
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2013-12; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Expressed Prostatic Secretions (EPS) for bacterial species in prostatitis patients vs controls | 1 day
  Expressed Prostatic Secretions (EPS) will be collected post Digital Rectal Exam (DRE). These biological samples will be tested for bacterial DNA rather than the traditional microbiological culturing techniques. Identification of these bacterial DNA will then be assessed between the groups to determine if prostatitis patients, in fact, do have more bacteria than normal controls.

SECONDARY OUTCOMES:
VB3 sample or first void after DRE for prostatitis patients vs controls | 1 day
  These biological samples will be tested for bacterial DNA rather than the traditional microbiological culturing techniques. Identification of these bacterial DNA will then be assessed between the groups to determine if prostatitis patients, in fact, do have more bacteria than normal controls.

OTHER OUTCOMES:
Chronic Prostatitis Symptom Index (CPSI) | 1 day
  Validated and standardized questionnaire for this area of research will be filled out by prostatitis patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No